CLINICAL TRIAL: NCT00694902
Title: A Single-centre, Randomized, Double-blind , Placebo Controlled, Dose Escalating Cross-over Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Inhaled Doses of GSK610677 and Placebo in Healthy Male Subjects
Brief Title: Single Dose Escalation Study FTIM in Order to Assess Safety and Tolerability of GSK610677
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: IP2107882
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Healthy Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Sequence 1 of Cohort-I (Experimental): Subjects in Sequence 1 will receive Placebo during treatment period 1, 50 microgram GSK610677 during treatment period 2 and 250 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 2 of Cohort-I (Experimental): Subjects in Sequence 2 will receive 10 microgram GSK610677 during treatment period 1, Placebo during treatment period 2 and 250 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 3 of Cohort-I (Experimental): Subjects in Sequence 3 will receive 10 microgram GSK610677 during treatment period 1, 50 microgram GSK610677 during treatment period 2 and Placebo during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 4 of Cohort-I (Experimental): Subjects in Sequence 4 will receive 10 microgram GSK610677 during treatment period 1, 50 microgram GSK610677 during treatment period 2 and 250 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677
- Sequence 5 of Cohort-II (Experimental): Subjects in Sequence 5 will receive Placebo during treatment period 1, 100 microgram GSK610677 during treatment period 2 and 500 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 6 of Cohort-II (Experimental): Subjects in Sequence 6 will receive 30 microgram GSK610677 during treatment period 1, Placebo during treatment period 2 and 500 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 7 of Cohort-II (Experimental): Subjects in Sequence 7 will receive 30 microgram GSK610677 during treatment period 1, 100 microgram GSK610677 during treatment period 2 and Placebo during treatment period 3.
  Interventions: Drug: GSK610677; Drug: Placebo
- Sequence 8 of Cohort-II (Experimental): Subjects in Sequence 7 will receive 30 microgram GSK610677 during treatment period 1, 100 microgram GSK610677 during treatment period 2 and 500 microgram GSK610677 during treatment period 3.
  Interventions: Drug: GSK610677
- Cohort III (Experimental): Subjects in Cohort III after randomization will either receive 1000 microgram GSK610677 or placebo.
  Interventions: Drug: GSK610677; Drug: Placebo

INTERVENTIONS:
Drug: GSK610677 — GSK610677 Multi-Dose Powder Inhaler will be available in the strength of 10, 50, 100 and 25 microgram with dose levels of 10, 30, 50, 100, 250, 500 and 1000 microgram. Subjects will receive GSK610677 as single inhale dose.
Drug: Placebo — Matching Placebo for GSK610677 will be available as Multi-Dose Powder Inhaler. Subjects will receive Placebo as single inhale dose.
  Arms: Cohort III; Sequence 1 of Cohort-I; Sequence 2 of Cohort-I; Sequence 3 of Cohort-I; Sequence 5 of Cohort-II; Sequence 6 of Cohort-II; Sequence 7 of Cohort-II

SUMMARY:
This study is the first administration of GSK610677 to man. The main aim of this clinical study is to investigate the safety and tolerability of different doses of the investigational medicinal product GSK610677. 2 cohorts of 8 subjects (Cohorts I and II) will be enrolled into this study. Individual subjects in each cohort will have up to 3 treatment periods. In each treatment period, subjects will receive a single inhaled dose of GSK610677 or placebo. Predicted doses are: 10, 30, 50 100 250 and 500ug.For individual subjects in each cohort, there will be a minimum wash out period of at least 10 days. In this period safety and tolerability data will be collected prior to dose to the next level.After safety review meetings between the site and the sponsor following the administration of the 500 ug dose, it was decided to add an extra cohort (Cohort III) of 8 subjects and administer 1000µg. Each subject in Cohort III will undergo a screening visit, one treatment period, and a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range and determined by the investigator to be of clinical significance for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with liver function values outside the normal range should always be excluded from enrolment.
* Male between 18 and 50 years of age.
* Subjects must agree to use one of the contraception methods listed in Section 8. This criterion must be followed from the time of the first dose of study medication until 7 days after the last dose of study medication or 5 terminal half-live after the last dose of the study medication, whichever is longer.
* Body weight > 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec.
* Demonstrated ability to use the DISKUS inhaler device in a satisfactory and repeatable manner as judged by the investigator or designee.
* Current non-smoker, who has not used any inhaled tobacco product in the 12 month period preceding the screening visit and who have a total pack history of < 5 pack years (pack years = (number of cigarettes per day/20) x (no. of years smoked)).
* Screening pre-bronchodilator FEV1 > 80% predicted and FEV1/FVC ratio > 0.7.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Subject is known to be HIV seropositive.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a half-pint (220 mL) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects who have asthma or a history of asthma.
* The subject has respiratory symptoms, including "cold or flu" type symptoms or any respiratory infection/symptoms within 4 weeks of screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits or grapefruit hybrids from 7 days prior to the first dose of study medication.
* Chronic liver or biliary disease, history of Gilbert's syndrome.
* History in increased liver function tests above upper limit of normal in the past six months.
* Subjects who are kept due to regulatory or judicial order in an institution.
* Subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05-26 (Actual); Primary Completion 2008-09-23 (Actual); Study Completion 2008-09-23 (Actual)

PRIMARY OUTCOMES:
Blood samples over a period of 48 hours. | Pre-dose, 5, 10, 15, 30 and 45 minutes, 1, 1.5, 2, 4, 6, 8, 12, 24 and 48 hours post dose

SECONDARY OUTCOMES:
Safety parameters over a period of the study, including ECG, Telemetry and vital sign. Continuous adverse event monitoring from dosing until study conclusion and follow up, 14-21 days after last dose. | Up to 21 days after last dose
Plasma GSK610677 and GSK1437357 concentrations | Up to 21 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study IP2107882 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/IP2107882?search=study&search_terms=IP2107882#rs